CLINICAL TRIAL: NCT01274936
Title: Effectiveness of a Compound Traditional Chinese Herbal Medicine, Qishe Pill, on Cervical Radiculopathy: a Randomized, Double-blind, Placebo-controlled, Multicentre Trial
Brief Title: Qishe Pill for Cervical Radiculopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Fudan University (Other); Changchun University of Chinese Medicine (Other); Lanzhou Hospital of Traditional Chinese Medicine (Other); Suzhou Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Cui xuejun, Vice director, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Qishe
Record Dates: First submitted 2010-12-14; First posted 2011-01-12 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — qishe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Qishe (Experimental)
  Interventions: Drug: Qishe Pill
- Control (Placebo Comparator): Qishe Placebo
  Interventions: Drug: Qishe Placebo

INTERVENTIONS:
Drug: Qishe Pill — Pill, 3.75 g, twice per day, four weeks
  Arms: Qishe
Drug: Qishe Placebo — Pill, 3.75 g, twice per day, four weeks
  Arms: Control

SUMMARY:
Radiculopathy generally presents with pain, numbness, or weakness in a dermatomal distribution. Cervical radiculopathy results from impingement on a nerve root by either spondylotic narrowing of the neural foramen or a lateral intervertebral disc herniation. Specifically, it should be the goal of the treating physician to relieve pain, improve function, and prevent recurrence. Various studies have shown that nonoperative management of cervical radiculopathy leaves a substantial minority of patients with persistently troublesome symptoms. Pharmacologic agents treat the underlying condition and provide symptomatic relief. The various classes of medications used to treat radiculopathy include steroids, nonsteroidal antiinflammatory drugs (NSAIDs), muscle relaxants, narcotics, and antidepressants. Herbal medicines have been used for centuries in China. In China, many patients with cervical disc disease are increasingly turning to herbal medicines to alleviate their symptoms and reduce the side effects of medications. The goal of this study is to determine the efficacy and efficacy of an herbal medicine, Qishe Pill, to treat cervical radiculopathy.

DETAILED DESCRIPTION:
Cervical radiculopathy is a distinct consideration in the evaluation of any patients who have neck pain and may be defined simply as an abnormality of a nerve root, which originates in the cervical spine. The initial approach to the management of cervical spondylopathy radiculopathy is nearly the same that the nonspecific neck or back pain can be found in most of patients. Conservative treatments include non-steroidal anti-inflammatory drugs (NSAIDs), narcotics, muscle relaxants, physical therapy and transcutaneous electrical nerve stimulation (TENS). The main objectives of conservative treatments are to relieve pain, improve function and improve health-related quality of life.However, these treatments for cervical radiculopathy are limited by their modest effectiveness. Surgical treatment for cervical disc disease is indicated when symptoms are refractory to conservative treatments and neurological symptoms are progressive. In terms of pharmacotherapy, there generally is no randomized, placebo-controlled trial available comparing the standard nonsurgical treatments. Therefore, care plans should be designed principally based on accumulated experience, the services available locally, and the respective preferences of patients. Treatment plans are developed to alleviate pain, improve function, and prevent recurrences.

As a complementary and alternative medicine (CAM), herbal medicines have the potential to avoid the adverse effects of medications and surgery.In the basic theory of traditional Chinese medicine (TCM), the obstruction of Qi flow and blood circulation in the neck area caused by some pathogenic factors, such as "Feng"(wind), "Han"(cold), "Shi"(dampness), invading the neck, induces cervical degenerative disc diseases which are the cause of cervical radiculopathy. According to the four traditional methods of diagnosis - observation, listening, interrogation, and pulse-taking, on patients, TCM doctors can analyze the certain pathogenic factors which cause neck pain. And then they will prescribe herbal formulae based on the effect and the main indications of Chinese medicine. Natural substances, including herbal medicines, have being used to promote healing and alleviate neck pain in western countries. Previous studies have demonstrated that some active substances in herbal medicine can promote Qi flow and blood circulation to alleviate pain.

A number of studies on the effects of the Chinese herbal medicine on cervical radiculopathy have been proposed, but useful empirical research is insufficiency. For chronic neck pain with or without radicular symptoms, there is low quality evidence that herbal is more effective than placebo for pain relief, which is measured at the end of the treatment. However, the size of the studies was small and the effect was measured in the short-term. Further research is very likely to change both the effect size and our confidence in the results. There is a need for trials with adequate numbers of participants that address long-term efficacy or effectiveness of herbal medicine compared to placebo.

Qishe Pill is composed of processed Radix Astragali, Muscone, Szechuan Lovage Rhizome, Radix Stephaniae Tetrandrae, Ovientvine, Calculus Bovis Artifactus. Using a well-designed clinical trial, we will survey the effectiveness of concurrent use of this remedy in relieving neck pain. Therefore, the present study is to examine effectiveness and safety of Qishe Pill, a compound traditional Chinese herbal medicine, on neck pain in cervical spondylotic radiculopathy in a randomized, double-blind, placebo-controlled trial. Results of this study will provide evidence regarding the value of the Qishe Pill as an intervention to alleviate neck pain caused by cervical radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of chronic neck pain since at least 3 months and complaints for a maximum duration of 5 years.
* average pain intensity of the last 7 days more or equal to 25 points measured by a Neck Disability Index.
* intellectual and physical ability to participate in the study.
* informed consent.
* One positive result of Brachial Plexus Traction Test, Cervical compression test or Cervical distraction test

Exclusion Criteria:

* cervical pain related to malignancy
* cervical pain due to an accident
* inflammatory joint disorders
* previous spine surgery
* protrusion/prolapse of a spinal disk, spondylolisthesis, with radicular symptomatology
* actually doing or planning to do other regular physical exercise during the study with possible positive effects on neck pain - such as swimming, yoga, pilates, tai chi, etc.
* use of pain drugs for other diseases (> 1x/week)
* pregnancy
* severe chronic or acute disease interfering with therapy attendance
* alcohol or substance abuse
* participation in another clinical trial in the last 6 months before study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-02 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
pain severity(measured with a visual analogue scale, VAS) | changes from baseline at 2 weeks
  Operationally, the VAS score display as a horizontal line, 100 mm in length, word descriptors anchored at each end. The patient marks on the line the point that they feel represents their perception of their current pain. The VAS score is then determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.
pain severity(measured with a visual analogue scale, VAS) | changes from baseline at 4 weeks
  Operationally, the VAS score display as a horizontal line, 100 mm in length, word descriptors anchored at each end. The patient marks on the line the point that they feel represents their perception of their current pain. The VAS score is then determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.

SECONDARY OUTCOMES:
SF-36 | changes from baseline at 2 weeks
  a composite of functional status
Neck Disability Index（NDI） | changes from baseline at 2 weeks
  a composite of functional status
Patient satisfaction degree | Changes from baseline at 4 weeks
  To evaluate satisfaction
SF-36 | changes from baseline at 4 weeks
  a composite of functional status
Neck Disability Index（NDI） | changes from baseline at 4 weeks
  a composite of functional status
Neck Disability Index（NDI） | changes from baseline at 3 months
  a composite of functional status
Neck Disability Index（NDI） | changes from baseline at 6 months
  a composite of functional status
Safety evaluation | changes from baseline at 4 weeks
  Safety evaluation
The medicine issue | changes from baseline at 2 weeks
Compliance assessment | changes from baseline at 2 weeks
  To evaluate compliance
Compliance assessment | changes from baseline at 4 weeks
  To evaluate compliance
Concomitant medication | changes from baseline at 2 weeks
Concomitant medication | changes from baseline at 4 weeks
X-ray(frontal and lateral) | changes from baseline at 4 weeks
Kidney function test | changes from baseline at 4 weeks
Liver function test | changes from baseline at 4 weeks
ECG | changes from baseline at 4 weeks
Occult Blood | changes from baseline at 4 weeks
Excrement routine | changes from baseline at 4 weeks
Urine routine | changes from baseline at 4 weeks
Blood routine | changes from baseline at 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Dr, Principal Investigator — Longhua Hospital
Locations (5):
- China (5):
  - No.1 Hospital, Changchun University of TCM, Changchun
  - Gansu Hospital of TCM, Lanzhou
  - Huadong Hospital, Shanghai
  - Longhua Hospital, Shanghai
  - Suzhou Hospital of TCM, Suzhou

REFERENCES:
- [Derived] Cui XJ, Sun YL, You SF, Mo W, Lu S, Shi Q, Wang YJ. Effects of Qishe Pill, a compound traditional Chinese herbal medicine, on cervical radiculopathy: study protocol for a randomized controlled trial. Trials. 2013 Oct 7;14:322. doi: 10.1186/1745-6215-14-322. PMID 24099350